CLINICAL TRIAL: NCT04685356
Title: Effect of the Infant Behavioral Assessment and Intervention Program (IBAIP) in Preterm Infants on Neurodevelopment at 2 Years Corrected Age
Brief Title: Effect of the IBAIP in Preterm Infants Neurodevelopment
Acronym: IBAIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 29BRC17.0219
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth | interventions — Glycation End Products, Advanced; Psychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IBAIP Group (Experimental): Children benefiting from assessment and intervention providing by a healthcare professional (physiotherapist or psychomotor therapist) trained and certified for IBAIP. This care will take place upon discharge from the hospital at the rate of one session per month for 6 months. The sessions will take place in the presence of at least one of the parents and at home. These children will also benefit from standard follow-up (medical follow-up, paramedical or specialized medical support depending on the development and needs).
  Interventions: Other: IBAIP : Infant Behaviour Assessment and Intervention Program; Other: Ages and Stages Questionnaire (ASQ); Other: Parenting Stress Index (PSI); Other: Bayley Scales of Infant and Toddler Development (BSID-IV)
- Control group (Active Comparator): Children benefiting from standard care upon discharge from hospital with 1 medical consultation per month and, medical sepcialist and / or paramedical(physiotherapy, speech therapy, psychomotricity, etc.). consultations if indicated by the physician providing follow-up
  Interventions: Other: Standard Support; Other: Ages and Stages Questionnaire (ASQ); Other: Parenting Stress Index (PSI); Other: Bayley Scales of Infant and Toddler Development (BSID-IV)

INTERVENTIONS:
Other: IBAIP : Infant Behaviour Assessment and Intervention Program — The IBAIP intervention program consists of providing an intervention with the child and their family, at home, upon discharge from hospital and up to a corrected age of 6 months. Interventions therefore take place at the early stage of the child's brain development. The intervention is performed by a IBAIP-trained and certified physiotherapist or psychomotor therapist trained , at the rate of one session per month over a period of approximately 6 to 8 months (6 months of corrected age). The session takes place in the child's usual living environment, at home, in the presence of at least one of the parents. It focuses on the child's behaviors and consists of assisting the family in its interactions with the child so that these are adapted and responsive to the child's development needs over time through repeated interventions.
  Arms: IBAIP Group
Other: Standard Support — One medical consultation per month and, if indicated by the physician providing follow-up, medical specialist and / or paramedical (physiotherapy, speech therapy, psychomotricity, etc.) consultations including interventions in the case of developmental delays
  Arms: Control group
Other: Ages and Stages Questionnaire (ASQ) — Global development screening tool
Other: Parenting Stress Index (PSI) — Index used to detect difficulties sufficiently significant that they might require psychosocial intervention
Other: Bayley Scales of Infant and Toddler Development (BSID-IV) — This test was designed to measure the development of infants / young children. This assessment examines all spheres of child development, identifies children with developmental delay and assesses children's developmental performance compared to their peers.

SUMMARY:
Mortality in very preterm infants has decreased significantly over the past twenty years. However, neuromotor, behavioral and cognitive development disorders are more common in these children born before 33 weeks of gestation as compared to term born infants.

These neurodevelopmental disorders include difficulties with self-regulation, tone, posture or poor quality movements as well as inadequate responses to sensory simulation.

Post-hospital discharge follow-up and interventionsof children born very preterm ares very heterogeneous in France. They are mainly carried out in a rehabilitation center, based on caregivers whereas IBAIP is carried out at home and family centered.

Early interventions during hospitalization or after discharge appear potentially of great interest in improving the neurodevelopemental outcome of the very preterm infants. Several early interventions have been developed and evaluated in other countries. These interventions are designed to be used early in life, mainly during the first 3 years of life, and are based on brain plasticity and intense synaptogenesis during this period of life.

The IBAIP (Infant Behavior Assessment and Intervention Program) was developed on the same theoretical foundations as the NIDCAP (Neonatal Individualized Development Care and Assessment Program). IBAIP consists of providing the child and his family with an intervention, at home, starting just before hospital discharge up to a 6 months corrected age. .The aim of IBAIP is to support developmental functions including infant's self-regulation and focus on improving the responsiveness of parents' infant interactions.

DETAILED DESCRIPTION:
This program consists of providing intervention, by a IBAIP trained and certified healthcare professional, with the child and his family, starting a few days before hospitalization discharge (hospital or home care) and continuing at home until the corrected age of 6 months. It focuses on the child's behaviors and consists of assisting the family in its interactions with the child so that these are adapted and responsive to the child's development needs over time through repeated interventions.

A cluster randomization will be used meaning the centers are randomized, not the individual patients. The centers will be randomized before the inclusion of patients in order to allow the physiotherapists or psychomotor therapists to be trained and certified to the IBAIP before the start of the trial.

Visit 1: Upon discharge from hospital, follow-up as part of standard care (control group) with at least 1 medical consultation per month during the first 6 months or according to the IBAIP program (experimental group) with one intervention before discharge from hospital and at home after hospital discharge, with1 session once a month up to 6 months corrected age (i.e. 6 to 8 sessions) in addition to standard care.

Visit 2: At 6 months corrected age, parents' response to the PSI (Parenting Stress Index) questionnaire.

Visit 3: At two years corrected age :

* Assessment of the development quotient obtained on the BSID-IV scale during a consultation with a neuro-psychologist or pediatrician.
* Parents' response to the PSI (Parenting Stress Index) questionnaire
* Parents' response to the ASQ (Ages and Stages Questionnaire

ELIGIBILITY:
Inclusion Criteria :

* Preterm infants born (including multiple pregnancies) at a gestational age between 25 weeks +0 days and 32 weeks + 6days.
* Written informed consent of at least one of the parents / legal guardian or 2 parents / legal guardians depending on the family context
* Normal neurological examination between 36 and 41 weeks of corrected age

Exclusion Criteria:

* Intraventricular hemorrhage (III or IV), periventricular leukomalacia
* Brain MRI abnormalities performed after 36 weeks of corrected age
* Life-threatening pathology
* Severe congenital abnomality
* Severe maternal pathology (physical and / or mental)
* Parents whose native languageis not French
* Participation in another interventional study on the management of post-hospital neurodevelopment disorders

Ages: 25 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2028-01-08 (Estimated); Study Completion 2028-01-08 (Estimated)

PRIMARY OUTCOMES:
To assess the effect of the Infant Behavior Assessment and Intervention Program Program (IBAIP) in very preterm infants (< 33 weeks of gestation) on neurodevelopment at the corrected age of 2 years | 2 years of corrected age
  Patient neurodevelopment will be assessed using the Bayley Scales of Infant and Toddler Development (BSID-IV) scale. This test studies the different notions of development: cognitive, language, motor skills, socio-emotional, behavioral, communication and autonomy.

SECONDARY OUTCOMES:
To assess the effect of IBAIP on the 5 sub-scores of BSID-IV: cognitive, language, motor, socio-emotional and behavioral adaptive | 2 years of corrected age
  The BSID-IV scale can be analyzed at the level of each of these subscales. The different scores obtained allow us to identify precisely at what level the effect on neurodevelopment was the most significant.
To assess the effect on the stress level of mothers and fathers | 2 years of corrected age
  To assess through the response to the Parental Stress Index. This questionnaire consists in 120 items using a 5-level Likert scale. It allows the assessment of life stress score, parental stress and child stress.
Parental assessment of psychomotor development | 2 years of corrected age
  Ages and Stages questionnaire completed by the parents to assess the child's neurodevelopment in 5 areas (fine motor skills, gross motor skills, communication, problem solving, individual or social skills).

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - CHU Angers, Angers
  - CHU Besançon, Besançon
  - CHU Brest, Brest
  - CHU Caen, Caen
  - CHU Grenoble, Grenoble
  - CHU Nantes, Nantes
  - CHU Rennes, Rennes
  - CHRU Strasbourg, Strasbourg
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Derived] Smith M, Kuhn P, Thiriez G, Debillon T, Datin-Dorriere V, Leboucher B, Mitanchez D, Courtois-Communier E, Sizun J, Roue JM. Infant behavioural assessment and intervention program to support neurodevelopmental outcome of very preterm infants at two years corrected age: a cluster randomised controlled trial study protocol. BMJ Open. 2025 Sep 4;15(9):e088167. doi: 10.1136/bmjopen-2024-088167. PMID 40908020